CLINICAL TRIAL: NCT04933630
Title: Tracking Response to Antidepressants in Advance of Investigational Trials, Relapse Study
Acronym: TRAIT-RS
Status: Completed | Type: Observational
Sponsor: Adams Clinical (Network)
Responsible Party: Sponsor
Other Study IDs: TRAIT-MDD-401
Record Dates: First submitted 2021-06-14; First posted 2021-06-22 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Selective Serotonin Reuptake Inhibitors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: FDA-approved selective-serotonin reuptake inhibitors (SSRIs) and selective-norepinephrine reuptake inhibitors (SNRIs) — Participants exiting the TRAIT study will have received a 90-day supply of their current protocol-approved antidepressant treatment (ADT) if clinically appropriate, prior to entering the TRAIT-RS study, in addition to a continuity of care letter to be given to their medical provider to facilitate a refill of that medication as desired. (See NCT04748276 for specific formulary and prescribing guidelines).

SUMMARY:
TRAIT-RS is an observational study to evaluate ongoing treatment response stability to standard of care antidepressant treatments (ADTs) among individuals who met criteria for Major Depressive Disorder (MDD) and completed the Tracking Response to Antidepressants in Advance of Investigational Trials (TRAIT) study (NCT04748276).

ELIGIBILITY:
Inclusion Criteria:

* Participant has completed the TRAIT study and, in the opinion of the investigator, would benefit from ongoing depression monitoring and/or ADT treatment.
* Participant has signed an ICF prior to any study-specific procedures being performed.
* Participant is male or female of age ≥ 18 years.
* Participant is in good physical health and, in the opinion of the investigator, is a suitable candidate for treatment with an ADT.

Exclusion Criteria:

* Participant is pregnant, breast-feeding, or planning to become pregnant.
* A history or presence of a clinically significant hepatic, renal, gastrointestinal, cardiovascular, endocrine, respiratory, immunologic, hematologic, dermatologic, or neurologic abnormality, which, in the opinion of the investigator, may impact participant safety or study results.
* Participant has a history of any psychiatric condition other than MDD, which, in the opinion of the investigator, is primary or any other psychiatric or neurologic disorder or symptom that could pose undue risk to the participant or compromise the study.
* Any participant who represents an acute suicidal risk in the opinion of the investigator.
* Moderate or severe substance use disorder within 90 days prior to screen according to DSM-5 criteria that, in the opinion of the investigator, could pose undue risk to the participant or compromise the study.
* Any condition that, in the opinion of the investigator, makes the participant unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults who previously met the Diagnostic and Statistical Manual - Version 5 (DSM-5) criteria for Major Depressive Disorder (MDD), sought enrollment in an industry-sponsored antidepressant trial, achieved MDD symptom remission in the TRAIT study, and, in the opinion of the investigator, would benefit from ongoing depression monitoring and/or ADT treatment.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2022-10-05 (Actual)

PRIMARY OUTCOMES:
Stability of treatment response as defined as change in self-report PHQ-9 total scores during the observational period from Baseline/Day 0 to End of Study (EOS)/Day 365. | Up to 52 weeks

SECONDARY OUTCOMES:
The number of participants who meet MDD relapse criteria as defined as the higher of a) PHQ-9 score ≥ 10, or b) ≥ 50% increase in PHQ-9 score from Baseline/Day 0, and verified by clinician-rated assessment as indicated by a HAM-D score ≥ 14 and CGI ≥ 4. | Up to 52 weeks
The number of participants who maintain ADT compliance as defined as ≥ 80% average monthly adherence during the observational period. | Up to 52 weeks

OTHER OUTCOMES:
The number of non-relapsing participants who elect to continue ADT treatment when incurring medication costs following an initial no-cost 90-day supply. | Up to 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jenicka Engler, PsyD, Principal Investigator — Adams Clinical
Locations (1):
- Adams Clinical, Watertown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided